CLINICAL TRIAL: NCT02374372
Title: Prospective Randomized Study Comparing the Hemodiafiltration On-line and Conventional Hemodialysis in Terms of Cost-benefit
Brief Title: Comparing the Hemodiafiltration On-line and Conventional Hemodialysis in Terms of Cost-benefit
Acronym: PHARMACO-$
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE10.253
Record Dates: First submitted 2013-09-24; First posted 2015-02-27 (Estimated); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Chronic Renal Failure; Hemodialysis
Keywords: hemodialysis; beta microglobulin; amyloidosis
MeSH Terms: conditions — Kidney Failure, Chronic; Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional hemodialysis (Active Comparator): conventional hemodialysis
  Interventions: Device: conventional hemodialysis
- hemodiafiltration On-line (Active Comparator): hemodiafiltration On-line
  Interventions: Device: hemodiafiltration On-line

INTERVENTIONS:
Device: conventional hemodialysis
  Arms: conventional hemodialysis
Device: hemodiafiltration On-line
  Arms: hemodiafiltration On-line

SUMMARY:
The site where the clinical trial will be conducted is at the St-Luc hospital from the CHUM. This is a prospective randomized study that will compare the two treatment modalities, HD and HDF, through economics and pharmaco-economics parameters.

Patients, who had previously been randomized in the CONTRAST study, will remain in their respective group and monitoring will continue. The next patients will be randomized in the same way (1: 1) using the same inclusion and exclusion criteria. HDF randomized patients will receive post-dilution standard reinjection (at least 100ml/min or 6 liter/hr). In rare cases, HDF patients can briefly have reinjection on a pre-dilution mode (if heparin need to be avoided for example) and the reinjection flow should be adjusted accordingly (200ml/min).

Length and frequency of sessions will be the same in the 2 groups. Blood tests will not change and will be the same than those used as routine assessments. Metabolic control of patients will be maintained according to the guidelines. Patients will be monitored for a minimum of 3 years. A set of demographic and clinical data will be collected from patient medical records and throughout the study.

Biochemical data as part of the usual blood tests of dialysis patients will be collected each month as well as will be stored and analyzed information about the annual cardiac ultrasounds.

All events will be scored (hospitalizations, patterns, duration) and the list and cost of drugs will be compiled every three months. These data will be useful in the economic analysis comparing the two treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years old,
* able to consent,
* patient needs to be on hemodialysis more than 8-12 hours a week (2-3 sessions)

Exclusion Criteria:

* severe none compliance (often missing sessions without good reasons),
* life expectation less than 3 months,
* treated with high-flux filters in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2011-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
compare the medication cost between the 2 groups (HD and HDF) | 3 years
demonstrate lower cost of erythropoietin in HDF, with same control of anemia to HD group | 3 years
demonstrate lower cost of phosphate binder in HDF, with same control of phospho calcium balance to HD group | 3 years

SECONDARY OUTCOMES:
demonstrate lower need of Erythropoietin and best control of anemia in HDF | 3 years
demonstrate lower need of phosphate binder and best control of phospho-calcique balance in HDF | 3 years
demonstrate less hospitalization stay and cost related in HDF group | 3 years
stabilisation or regression of left ventricular hypertrophy | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier Universitaire de Montréal (CHUM), Montreal, Quebec, Canada